CLINICAL TRIAL: NCT05329324
Title: Evaluation of Neuropathic Pain in Lipedema
Brief Title: Is The Pain in Lipedema Patients Neuropathic Pain?
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nihan ERDINC GUNDUZ, MD, Dokuz Eylul University
Other Study IDs: İzellipodemTez
Record Dates: First submitted 2022-04-04; First posted 2022-04-15 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema | interventions — Surveys and Questionnaires; Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group - Lipedema: Questionnaire for study group
  Interventions: Other: Questionnaire for study group
- Control Group - Acute Subacromial Impingement: Questionnaire for control group
  Interventions: Other: Questionnaire for control group

INTERVENTIONS:
Other: Questionnaire for study group — Demographic features, Stage and Type, The LANSS Pain Scale and Pain Detect Questionnaire to assess patients' pain characteristics,the Nottingham Health Profile to assess quality of life, and the Hospital Anxiety and Depression Scale to detect the presence of depression and anxiety will be completed by patients.
  Groups: Study Group - Lipedema
Other: Questionnaire for control group — Demographic features, The LANSS Pain Scale and Pain Detect Questionnaire to assess patients' pain characteristics,the Nottingham Health Profile to assess quality of life, and the Hospital Anxiety and Depression Scale to detect the presence of depression and anxiety will be completed by patients.
  Groups: Control Group - Acute Subacromial Impingement

SUMMARY:
Lipedema is a chronic progressive disease characterized by abnormal increase of subcutaneous adipose tissue. It is characterized by bilateral enlargement of the lower and/or upper extremities, typically sparing the hands and feet. This disease, which almost always affects women, has rarely been described in men due to hormonal disorders or concomitant diseases such as cirrhosis. Although the results vary, it has been reported that it is seen at a minimum rate of 1:72.000 or 11% of women are affected by this disease. Although it is a common disease, it can often be missed in daily practice. Therefore, it is very important to define the disease clinic well. Lipedema usually presents with swelling in the bilateral extremities. It begins in the post-adolescent period and is progressive. It does not respond to diet and exercise, does not improve with elevation, is spontaneous or painful to touch. Patients describe easy bruising with touch or minor trauma. In early lipedema, pain may be the main complaint in the extremities before the development of skin findings. Because of the absence of a defined clear pain pattern in these patients, diagnosis can be missed and confused with other diseases. In addition, it causes limitations in treatment of the pain. Adipose tissue can cause nociceptive and neuropathic pain because it contains both nociceptive neurons and neural innervation. It isn't known whether lipedema pain is of nociceptive or neuropathic origin. In different studies, the pain pattern is defined in different ways such as hyperalgesia, allodynia, spontaneous pain, blunt, heaviness, pressure, tearing, stabbing, severe and unbearable. In this study, the investigators aim to determine if the pain characteristics of patients with lipedema is neuropathic or not and to define the pain characteristics better in order to ensure earlier recognition and treatment of pain.

DETAILED DESCRIPTION:
This study is a descriptive cross-sectional study. 42 patients will be included to study who apply to the outpatient clinic of Dokuz Eylul University Faculty of Medicine, Department of Physical Therapy and Rehabilitation, and who are diagnosed or followed up with the diagnosis of lipoedema, aged between 18- 65 years. For the control group, 42 patients who had shoulder pain for less than 3 months and is diagnosed with acute subacromial impingement will be included as the nociceptive pain model. The LANSS Pain Scale and Pain Detect Questionnaire to assess patients' pain characteristics, the Nottingham Health Profile to assess quality of life, and the Hospital Anxiety and Depression Scale to detect the presence of depression and anxiety will be completed by patients. LANSS Pain Scale is an evaluation form that helps to understand whether the nerves carrying pain signals are working normally, and it consists of two parts, including a pain questionnaire and a sensory evaluation. As a result of the calculation made according to answers, a score above 12 is associated with the presence of neuropathic pain. Pain Detect Questionnaire consists of questions about characteristics, severity and spread of the pain, and it provides the opportunity to score with 5 options as none, very mild, mild, moderate, severe, very severe. This survey, which consists of 38 points in total; in the presence of above 19 points, the neuropathic pain component is interpreted as possible. Nottingham Health Profile consists of 6 sections and a total of 38 questions evaluating patients' pain, emotional reaction, sleep, social isolation, physical activity and energy. In this questionnaire, where the highest score is 600 points, a high score is associated with a deterioration in quality of life. Hospital Anxiety and Depression Scale consists of 14 questions about anxiety and depression and 4 options for each question. According to the results, 0-7 points were interpreted as normal, 8-10 points were considered borderline, and 11 points and above were interpreted as abnormal. According to results of questionnaires, the datas will be compared with statistical analysis. As a result, the investigators aim to say that lipedema pain is or is not a neurpathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-65
* Diagnosed with lipoedema
* Those who agreed to participate in the study
* To be at the appropriate sociocultural level to participate in the study
* For the control group, the patient has a diagnosis of acute subacromial impingement syndrome

Exclusion Criteria:

* Having type 1 or type 2 diabetes
* Patients with uncontrolled thyroid dysfunction
* Patients with chronic venous insufficiency and/or lymphedema
* Patients with acute or chronic renal failure
* Heart failure
* Having cancer or continuing cancer treatment
* Diagnosed with polyneuropathy
* Those with radiculopathy
* Patients with advanced degenerative joint disease in the affected extremity
* Those who have received antiepileptic, antidepressant medication in the last 6 months
* Persons with visual and hearing impairments that impair adaptation to work
* Patients who are illiterate and have cognitive impairment that will prevent them from giving written consent will not be included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 42 patients will be included to study who apply to the outpatient clinic of Dokuz Eylul University Faculty of Medicine, Department of Physical Therapy and Rehabilitation, and who are diagnosed or followed up with the diagnosis of lipoedema, aged between 18- 65 years. For the control group, 42 patients who had shoulder pain for less than 3 months and is diagnosed with acute subacromial impingement will be included as the nociceptive pain model.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
LANSS Pain Scale | Baseline
  LANSS Pain Scale is an evaluation form that helps to understand whether the nerves carrying pain signals are working normally, and it consists of two parts, including a pain questionnaire and a sensory evaluation. As a result of the calculation made according to answers, a score above 12 is associated with the presence of neuropathic pain.
Pain Detect Questionnaire | Baseline
  Pain Detect Questionnaire consists of questions about characteristics, severity and spread of the pain, and it provides the opportunity to score with 5 options as none, very mild, mild, moderate, severe, very severe. This survey, which consists of 38 points in total; in the presence of above 19 points, the neuropathic pain component is interpreted as possible

SECONDARY OUTCOMES:
Nottingham Health Profile | Baseline
  Nottingham Health Profile consists of 6 sections and a total of 38 questions evaluating patients' pain, emotional reaction, sleep, social isolation, physical activity and energy. In this questionnaire, where the highest score is 600 points, a high score is associated with a deterioration in quality of life
Hospital Anxiety and Depression Scale | Baseline
  Hospital Anxiety and Depression Scale consists of 14 questions about anxiety and depression and 4 options for each question. According to the results, 0-7 points were interpreted as normal, 8-10 points were considered borderline, and 11 points and above were interpreted as abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Ebru sahin, MD, Study Director — Dokuz EU
Locations (1):
- Dokuz Eylul Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WOLD LE, HINES EA Jr, ALLEN EV. Lipedema of the legs; a syndrome characterized by fat legs and edema. Ann Intern Med. 1951 May;34(5):1243-50. doi: 10.7326/0003-4819-34-5-1243. No abstract available. PMID 14830102
- [Background] Akçalı Y, Atabey R. Lipödem ve Lipolenfödem: Tanı ve Tedavi, Türkiye Klinikleri J Cardiovasc Surg-Special Topics. 2018; 10:56-72
- [Background] Herbst KL, Mirkovskaya L, Bharhagava A, Chava Y, T. Te CH. Lipedema Fat and Signs and Symptoms of Illness, Increase with Advencing Stage, Archives of Medicine. 2015; 7:1-8
- [Background] Torre YS, Wadeea R, Rosas V, Herbst KL. Lipedema: friend and foe. Horm Mol Biol Clin Investig. 2018 Mar 9;33(1):/j/hmbci.2018.33.issue-1/hmbci-2017-0076/hmbci-2017-0076.xml. doi: 10.1515/hmbci-2017-0076. PMID 29522416
- [Background] Child AH, Gordon KD, Sharpe P, Brice G, Ostergaard P, Jeffery S, Mortimer PS. Lipedema: an inherited condition. Am J Med Genet A. 2010 Apr;152A(4):970-6. doi: 10.1002/ajmg.a.33313. PMID 20358611
- [Background] Szel E, Kemeny L, Groma G, Szolnoky G. Pathophysiological dilemmas of lipedema. Med Hypotheses. 2014 Nov;83(5):599-606. doi: 10.1016/j.mehy.2014.08.011. Epub 2014 Aug 23. PMID 25200646
- [Background] Ayhan FF. Lipödem: Klinik Tanı, Evreleme, Tiplendirme, Değerlendirme ve Tanı Kriterleri.Tanıdan Tedaviye Lipödem Sağlık Profesyonelleri İçin Rehber Kitap. Borman P, Dalyan M, Figen Ayhan FF eds. Hipokrat Kitabevi, Ankara 2019:17-34
- [Background] Aksoy H, Karadag AS, Wollina U. Cause and management of lipedema-associated pain. Dermatol Ther. 2021 Jan;34(1):e14364. doi: 10.1111/dth.14364. Epub 2020 Oct 12. PMID 33001552
- [Background] Angst F, Benz T, Lehmann S, Sandor P, Wagner S. Common and Contrasting Characteristics of the Chronic Soft-Tissue Pain Conditions Fibromyalgia and Lipedema. J Pain Res. 2021 Sep 17;14:2931-2941. doi: 10.2147/JPR.S315736. eCollection 2021. PMID 34557035
- [Background] Shavit E, Wollina U, Alavi A. Lipoedema is not lymphoedema: A review of current literature. Int Wound J. 2018 Dec;15(6):921-928. doi: 10.1111/iwj.12949. Epub 2018 Jun 29. PMID 29956468
- [Background] Yucel A, Senocak M, Kocasoy Orhan E, Cimen A, Ertas M. Results of the Leeds assessment of neuropathic symptoms and signs pain scale in Turkey: a validation study. J Pain. 2004 Oct;5(8):427-32. doi: 10.1016/j.jpain.2004.07.001. PMID 15501424
- [Background] Alkan H, Ardic F, Erdogan C, Sahin F, Sarsan A, Findikoglu G. Turkish version of the painDETECT questionnaire in the assessment of neuropathic pain: a validity and reliability study. Pain Med. 2013 Dec;14(12):1933-43. doi: 10.1111/pme.12222. Epub 2013 Aug 7. PMID 23924395
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Ömer A, Güvenir T, Küey, L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlilik ve Güvenilirlik Çalışması. Türk Psikiyatri Dergisi. 1997; 8: 280- 287.